CLINICAL TRIAL: NCT05280652
Title: N-CHEFS (Nutritional and Culinary Habits to Empower Families Towards Sustainability) - a Multicentric Pilot Study
Brief Title: Nutritional and Culinary Habits to Empower Families Towards Sustainability - a Multicentric Pilot Study
Acronym: n-CHEFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021.124
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Family Research
Keywords: culinary medicine; home cooking; family-based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Family intervention group (Experimental): Families (dyads parent and child) will attend culinary-nutritional workshops with theoretical and practical nutritional and culinary information (knowledge and skills to prepare healthy and easy menus) to follow a sustainable Mediterranean diet.
  Interventions: Behavioral: Nutritional and culinary intervention
- Parent-only intervention group (Experimental): Parents will attend culinary-nutritional workshops with theoretical and practical nutritional and culinary information (knowledge and skills to prepare healthy and easy menus) to follow a sustainable Mediterranean diet.
  Interventions: Behavioral: Nutritional and culinary intervention
- Control (Active Comparator): Families (dyads parent and child) will attend nutritional workshops with theoretical information to follow a sustainable Mediterranean diet.
  Interventions: Behavioral: Nutritional intervention

INTERVENTIONS:
Behavioral: Nutritional and culinary intervention — Participants will attend 6 two-hours nutritional-culinary workshops between May 2022 and February 2023. All of the workshops will be held in a kitchen, and will be given in groups of 2 dyads or parents according to the intervention group. In addition, during the intervention families will be given access to a web page with nutrition and culinary education materials (infographics, videos).
  Arms: Family intervention group; Parent-only intervention group
Behavioral: Nutritional intervention — Participants will attend 6 1-hour nutritional workshops between May 2022 and February 2023. The workshops will be held in person, and will be given in groups of 10-12 families. In addition, during the intervention families will be given access to a web page with nutrition education materials (infographics, videos).
  Arms: Control

SUMMARY:
Background: Different studies have shown that nutritional interventions can be effective in informing and educating the population about the need to follow a healthy diet to prevent obesity and other chronic diseases. However, sometimes this knowledge is difficult to apply in daily life, which is usually marked by lack of time and easy access to food alternatives that are not healthy but can be more comfortable. These difficulties may be greater in families today since the lack of time is greater and it is a greater challenge to get minors to consume a high amount (5 servings a day) of fruits and vegetables. Culinary medicine is an emerging discipline that combines nutrition and gastronomy to increase the prevention and treatment of chronic diseases.

Objective: The main objective is to demonstrate whether a culinary-nutritional intervention in families reduces the risk of obesity and increases adherence to a healthy and sustainable diet.

Methods: The present project will cover culinary medicine and home-cooking as innovative strategies to improve the eating habits of families through an intervention based on face-to-face nutricional-culinary workshops and online material, where apart from receiving nutritional education, they will be taught a series of culinary techniques (adapted to adults and children) so that they learn to cook in an easy, enjoyable and family-friendly way, with tools to eat healthier in a simple and quick way.

The intervention will be carried out with 92 families (dyads 1 adult and 1 child) which will be randomized in a 1: 1: 2 ratio into three groups: group 1 (intervention with families) in which families will attend nutritional-culinary workshops with theoretical and practical information to follow a sustainable Mediterranean diet; group 2 (intervention with parents) in which only parents will attend nutritional-culinary workshops with theoretical and practical information to follow a sustainable Mediterranean diet; and group 3 (control) in which families will attend nutritional workshops with theoretical information to follow a sustainable Mediterranean diet.

UPDATED NOTE AFTER RECRUITMENT: Due to financial and recruitment issues, a total of 29 families were recruited.

DETAILED DESCRIPTION:
The present pilot study is a multicentric study which will be carried out in two cities of Spain, Alicante and Madrid.

The study is divided into two periods: the 10-month intervention period and the 4-month follow-up period. The intervention period will be from May 2022 to February 2023 and the follow-up period from March 2023 to June 2023.

A total of 92 families will be included in the present study which will be randomized in a 1: 1: 2 ratio into three groups: group 1 (intervention with families) in which families will attend nutritional-culinary workshops with theoretical and practical information to follow a sustainable Mediterranean diet; group 2 (intervention with parents) in which only parents will attend nutritional-culinary workshops with theoretical and practical information to follow a sustainable Mediterranean diet; and group 3 (control) in which families will attend nutritional workshops with theoretical information to follow a sustainable Mediterranean diet.

The sample size was calculated according to the the results on the change in BMI between subjects who followed a culinary intervention vs subjects in the control group of the study by Gatto et al. (2017) (doi:10.1111/ijpo.12102). A sample size of 83 families (55 intervention group families, 28 control group families) was estimated to find a change between groups (intervention vs. control) in the z-score BMI of 0.06 points with a standard deviation (SD) of 0.09 points, with a power of 80% and an alpha error of 5%. Assuming a 10% dropout rate, the initial number of families recruited is increased to 92 (30-31 families in each of the three groups).

UPDATED NOTE AFTER RECRUITMENT: Due to financial and recruitment issues, a total of 29 families were recruited.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between 9-14 years old.
* The child is at risk of obesity because it is over cut-offs of BMI according to their age or because it has a low level of adherence to the Mediterranean dietary pattern (an score ≤7 points in the Kidmed questionnaire).
* There is at least 1 obesity risk factor in the household: one or both progenitors has overweight or obesity; one of both progenitors has only primary studies; one or both progenitors are unskilled workers; the total household number is ≤3; the child birthweight was >4 kg; biological mother smoked during pregnancy; biological mother's weight gain during pregnancy was greater than the cut-offs of weight according to her BMI before pregnancy; biological mother's BMI before pregnancy was ≥30 kg/m2; one or both progenitors has a low adherence to the Mediterranean diet (17 points Mediterranean diet score ≤8); or the score for the family nutrition and physical activity screening tool is ≤50.

Exclusion Criteria:

* The participant progenitor or child has any food allergies and intolerances incompatible with the Mediterranean diet (fruits, nuts).
* The participant progenitor or child follow a specific dietary pattern incompatible with the intervention.
* The participant progenitor or child has type 1 diabetes, severe diseases of the digestive system, kidney, cancer, other diseases that limit survival less than 1 year, or eating disorders.
* The family has not access to a PC, tablet or telephone with internet.
* The family has participated in cooking workshops in the past 3 years.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Effect of the intervention on changes in body mass index (BMI) | At baseline, and 10 and 14 months follow-up
  Weight will be measured with a Tanita RD-545 (Tanita Corp Tokyo Japan). Height will be measured to the nearest 0.1 cm using a portable stadiometer. Differences between intervention groups on changes on BMI between baseline and 10-months and baseline and 14-months follow up.

SECONDARY OUTCOMES:
Effect of the intervention on home cooking habits | At baseline, and 10 and 14 months follow-up
  A validated questionnaire will be used to assess the use of different culinary techniques (Culinary Habits Frequency Questionnaire). Differences between intervention groups on changes on culinary habits between baseline and 10-months and baseline and 14-months follow up.
Effect of the intervention on the adherence to the Mediterranean Diet (MedDiet) | At baseline, and 10 and 14 months follow-up
  Adherence to the MedDiet will be measured with the validated 17-item Mediterranean Diet Adherence questionnaire among aduls and the Kidmed questionnaire among children. Differences between intervention groups on changes on Mediterranean diet adherence between baseline and 10-months and baseline and 14-months follow up.
Home cooking attitudes and self-confidence on cooking at home with the cooking attitudes and self-confidence questionnaire | At baseline, and 10 and 14 months follow-up
  A non-validated questionnaire that measures cooking attitudes and self-confidence will be used at baseline and after 10-months of follow-up. The "cooking self-confidence and attitudes questionnaire" includes 18 questions on self-confidence and 18 questions on attitudes. Each question includes a 5-item Likert scale answer. A higher score means a higher self-confidence or positive attitude on home cooking.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - University of Navarra, Pamplona, Navarre
  - Universidad de Alicante, Alicante

REFERENCES:
- [Background] Enright G, Allman-Farinelli M, Redfern J. Effectiveness of Family-Based Behavior Change Interventions on Obesity-Related Behavior Change in Children: A Realist Synthesis. Int J Environ Res Public Health. 2020 Jun 8;17(11):4099. doi: 10.3390/ijerph17114099. PMID 32521815
- [Background] Smith JD, Montano Z, Dishion TJ, Shaw DS, Wilson MN. Preventing weight gain and obesity: indirect effects of the family check-up in early childhood. Prev Sci. 2015 Apr;16(3):408-19. doi: 10.1007/s11121-014-0505-z. PMID 25263212